CLINICAL TRIAL: NCT06857292
Title: Clinical Study on the Safety, Efficacy and Pharmacokinetics of Telpegfilgrastim Injection in Pediatric Cancer Patients with Chemotherapy
Brief Title: Clinical Study on the Safety, Efficacy and Pharmacokinetics of Telpegfilgrastim in Pediatric Cancer Patients with Chemotherapy
Acronym: Telpegfilgrast
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Telpegfilgrastim
Record Dates: First submitted 2024-12-02; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-Induced Neutropenia
Keywords: Telpegfilgrastim; pediatric cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Use Telpegfilgrastim to prevent chemotherapy-induced neutropenia
  Interventions: Drug: Telpegfilgrastim

INTERVENTIONS:
Drug: Telpegfilgrastim — Experimental group: Patients were subcutaneously injected with Telpegfilgrastim 33μg/kg (maximum dose ≤2mg) 24h after chemotherapy, 21 days for one chemotherapy cycle, and only one chemotherapy cycle was observed.
  Pharmacokinetic determination: Among them, 8 patients underwent pharmacokinetic determination. The pharmacokinetic sampling time points were blood samples taken before administration, 12 h, 24 h, 48 h, 120h, 168 h, 336 h, 480h after administration. A total of 8 blood samples were collected, and the pharmacokinetic characteristics of the experimental drugs were analyzed by ELISA.

SUMMARY:
This study is a multicenter, single-arm, prospective study. The study population includes children with cancer who require high-intensity chemotherapy. The study aims to evaluate the safety and effectiveness of Telpegfilgrastim in preventing neutropenia in children with cancer (neuroblastoma, sarcoma, lymphoma, etc.) undergoing chemotherapy, while also studying the pharmacokinetic characteristics of Telpegfilgrastim in children with cancer.

DETAILED DESCRIPTION:
Compared with the currently available straight chain PEG-rhG-CSF, the structure of its Y-type branch chain affects the activity and metabolic rate of the drug to a certain extent. While prolonging the half-life of the drug, the dosage of the drug is also significantly lower than that of the long-acting products on the market. It can be prophylactically administered once after chemotherapy to maintain the effective blood concentration of the whole cycle and effectively prevent the occurrence of neutropenia. Due to the reduction of the dose, the incidence of side effects such as musculoskeletal pain is correspondingly reduced, and there may be a better safety. At the same time, the accessibility of clinical PEG-rhG-CSF can be further solved, and the treatment cost is also expected to decrease, so that more patients can benefit from PEG-rhG-CSF.

Telpegfilgrastim was approved on June 30, 2023 for "reducing the incidence of infection characterized by febrile neutropenia in patients with non-myeloid malignants who are treated with myelosuppressive anticancer agents that tend to cause clinically significant febrile neutropenia." At present, although Telpegfilgrastim has been approved for neutropenia induced by chemotherapy for non-myeloid malignant tumors, the safety and efficacy data in pediatric patients are lacking, and the pharmacokinetic characteristics in children are still unclear. The aim of this study was to evaluate the safety and efficacy of Telpegfilgrastim in the prevention of neutropenia in pediatric cancer patients receiving chemotherapy, and to investigate the pharmacokinetics of Telpegfilgrastim in pediatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 14≤ age < 18 years;

  * Newly diagnosed patients with non-myeloid malignancies who are confirmed by histopathology or cytology to require intensive chemotherapy (first course of chemotherapy or second course of chemotherapy);

    * Primary prevention (G-CSF 24 to 72 hours after the first use of chemotherapy agents with myelosuppression to prevent the occurrence of febrile neutropenia (FN)) or secondary prevention (if FN or dose-restricted neutropenia occurred in a patient during a previous chemotherapy cycle) is required. Prophylactic use of G-CSF can be considered for the next chemotherapy cycle.

Febrile neutropenia (FN) : Oral temperature >38.3 ° C (axillary temperature >38.1 ° C) or oral temperature >38.0 ° C (axillary temperature >37.8 ° C) with ANC<0.5×10^9/L for 2 consecutive measurements within 2 hours, or ANC is expected to decrease to <0.5×10^9/L within 48 hours.

* KPS score ≥50 or Lansky (LPS) score ≥50;

  * Normal hematopoietic function of bone marrow (ANC≥1.5×10^9/L, PLT≥80×10^9 /L, Hb≥75g/L, WBC≥3.0×10^9/L, and not exceeding the upper limit of normal value);

    * Life expectancy of at least 6 months; ⑦ Obtain written informed consent.

Exclusion Criteria:

* Received any rhG-CSF within 3 weeks prior to study participation;

  * Received any antibody coupling drug (ADC) drugs with potential blood toxicity within 3 weeks before participating in the study;

    * Recipients of hematopoietic stem cell transplantation or organ transplantation;

      * Clinical trials of other drugs were being conducted within 2 months before enrollment;

        * There is no control of infection, body temperature ≥38℃; ⑥ Liver function test: total bilirubin (TBIL) alanine aminotransferase (ALT.) and aspartate aminotransferase (AST.) were more than 2.5 times the upper limit of normal value; ⑦ Renal function test: serum creatinine (Cr.) > 1.5 times the upper limit of normal value; ⑧Other conditions considered by the researchers to be contraindications for this study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall incidence of adverse reactions | 1 year
  The overall incidence of adverse reactions after prophylactic drug use during this period

SECONDARY OUTCOMES:
Incidence of grade 3-4 neutropenia | 3 weeks
  Incidence of grade 3-4 neutropenia during this period after prophylactic administration
Incidence of febrile neutropenia (FN) | 3 weeks
  Incidence of febrile neutropenia (FN) in this period after prophylaxis

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided